CLINICAL TRIAL: NCT04765319
Title: Delivery Considerations of Cognitive Processing Therapy for PTSD
Status: Completed | Type: Observational
Sponsor: VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Harrison R Weinstein, Principal Invesigator, VA Salt Lake City Health Care System
Other Study IDs: IRB_00133139
Record Dates: First submitted 2021-02-11; First posted 2021-02-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2021-02

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Vets: Veterans receiving care from the PTSD Clinical Team at the Salt Lake City VAMC. All participants are adults with a diagnosis of PTSD. This study plans on reviewing data collected as part of standard clinical practices. The study will have no impact on the treatment provided to the patient.
  Interventions: Behavioral: CPT for PTSD

INTERVENTIONS:
Behavioral: CPT for PTSD — Evidence based psychotherapy for PTSD

SUMMARY:
Review treatment outcomes of modifications to standard delivery of CPT for PTSD that are delivered as routine care at in VA outpatient clinic.

DETAILED DESCRIPTION:
Background and Introduction Cognitive Processing Therapy (CPT) is an evidenced based psychotherapy for PTSD. It is considered a first line treatment and has ample evidence supporting it's effectiveness (ISTSS and VA/DOD clinical practice guidelines). This therapy is manualized and a framework is provided to ensure consistent delivery. Additionally, the VA Office of Mental Health Operations sponsors training and dissemination of CPT throughout the VA system and the PI of this study is a trainer and consultant of this therapy. Flexibility exists in the protocol and CPT can be delivered in unorthodox modalities such as telehealth (Moreland et al, 2015) and on compressed time schedules (Held et al, 2020; Bryan et al, 2018). While the literature supports the effectiveness of these interventions in unique settings, no known studies have looked at outcome data of real-world outpatient clinics. The PTSD Clinical Team provides CPT as part of it's standard care with a variety of adaptations. The team practices measurement based care and routinely collects self-report symptom inventories to track patient progress. This study aims to use data collected as part of standard care in this clinic to evaluate the effectiveness of these treatment adaptations in this setting.

Purpose and Objectives The purpose of this study is to explore the impact of how CPT for PTSD is delivered. Initial areas of review will include in person vs. telehealth delivery and timing (daily vs. weekly).

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis
* Veterans eligible for VA care
* Treatment seeking Veterans

Exclusion Criteria:

* PTSD not priority of treatment due to comorbidity, safety, etc. All patients that would be treated for PTSD in outpatient clinic are included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans seeking treatment for PTSD at VA outpatient specialty clinic.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist 5 | Through study completion, an average of 12 sessions (3 months)
  Self report PTSD symptom inventory

SECONDARY OUTCOMES:
PHQ-9 | Through study completion, an average of 12 sessions (3 months)
  Self report depression symptom inventory

CONTACTS AND LOCATIONS:
Overall Officials: Harrison R Weinstein, PhD, Principal Investigator — VA Salt Lake City
Locations (1):
- Salt Lake City VAMC, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Not included in current IRB.